CLINICAL TRIAL: NCT02690441
Title: Physical Exercise Augmented Cognitive Behaviour Therapy for Older Adults With Generalised Anxiety Disorder
Brief Title: Physical Exercise Augmented CBT for GAD
Acronym: PEXACOG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solli Distriktspsykiatriske Senter (Other)
Collaborators: University of Bergen (Other); Norwegian University of Science and Technology (Other); University of Oslo (Other); University of California, Berkeley (Other); William Paterson University of New Jersey (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 971427272T1
Record Dates: First submitted 2016-02-05; First posted 2016-02-24 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: GAD; CBT; Physical exercise; Older adults
MeSH Terms: conditions — Generalized Anxiety Disorder; Motor Activity | interventions — Cognitive Behavioral Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT augmented with physical exercise (Experimental): Patients receive 10 sessions of cognitive behavioural therapy for generalized anxiety disorder. Patients also receive 5 weeks of physical exercise pre-treatment, and 10 weeks of physical exercise alongside CBT. Both treatment and physical exercise is administered individually.
  Interventions: Behavioral: Cognitive Behavioural Therapy; Behavioral: Physical Exercise
- CBT and placebo control (Active Comparator): Patients receive 10 sessions of cognitive behavioural therapy for generalized anxiety disorder. Patients also receive 5 weeks of placebo control (15 minutes telephone follow-up call each week) pre-treatment, and 10 weeks of attention placebo alongside CBT. Both treatment and placebo control is administered individually.
  Interventions: Behavioral: Cognitive Behavioural Therapy; Behavioral: Placebo control

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Cognitive behavioural therapy conducted individually. 10 weekly sessions, first session lasts 90 minutes, the remaining sessions last 45 minutes.
Behavioral: Physical Exercise — Manualised exercise. 15 weekly sessions with instructor, and two weekly unsupervised sessions performed individually.
  Arms: CBT augmented with physical exercise
Behavioral: Placebo control — One follow-up telephone call à 15 minutes each week for 15 weeks. Aims to control for therapist contact in physical exercise condition and total duration of treatment.
  Other Names: Telephone follow-up
  Arms: CBT and placebo control

SUMMARY:
Generalised anxiety disorder (GAD) is a severe and debilitating anxiety disorder that is highly prevalent among older adults. Anxiety and GAD is a well-documented risk factor for the development of other severe conditions such as depression and dementia, and effective treatments are called for. However, recommended treatment for GAD has consistently been found to yield blunted response rates for older adults compared to younger patients.

The purpose of this study is to evaluate the effects of exercise-augmented cognitive behaviour therapy for older adults with GAD. Exercise augmented CBT is expected to yield better results than standard CBT in terms of greater reduction of symptoms and increased rates of remission. The investigators will also investigate the effects of treatment on biological, physiological and neuropsychological measures.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of GAD

Exclusion Criteria:

* Substance abuse
* Use of benzodiazepines, use of antipsychotica
* Lack of ability to stabilize other psychotropic medication during participating in the study
* Medical condition that precludes participation in physical exercise
* Severe major depression as determined by the MINI International Neuropsychiatric Interview
* Life-time history of psychosis and/or mania
* Participation in other ongoing psychotherapy
* Organic brain disease
* Positive screening for dementia with Mini Mental State Examination
* Currently engaged in a regular physical exercise program

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2023-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in The Penn State Worry Questionnaire | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
  Assesses symptom severity of GAD
Change in clinical diagnosis after treatment assessed by independent, blinded rater with Anxiety Disorders Interview Schedule (ADIS-IV) | Baseline and post-treatment (up to 20 weeks after baseline)
  Remission rates. Assessed by independent, blinded rater with Anxiety Disorders Interview Schedule (ADIS-IV)

SECONDARY OUTCOMES:
Geriatric Anxiety Inventory | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
Generalized Anxiety Disorder 7-item scale (GAD-7) | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
Beck Anxiety Inventory | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
Beck Depression Inventory - II | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
Bergen Insomnia Scale | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
Quality of Life Inventory | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
International Physical Activity Questionnaire (IPAQ) | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
5-item Treatment Credibility and Expectancy Scale (CES) | Baseline

OTHER OUTCOMES:
Function and structure of prefrontal lobes and limbic system | Baseline, post-treatment (up to 20 weeks after baseline) and 12 months follow-up
  Functional Magnetic Resonance Imaging (fMRI) conducted with a 3-Tesla scanner.
Blood samples | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
  Serum concentrations of mature and pro brain-derived neurotropic factor
Saliva samples | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
  To measure cortisol
Three subtests from Delis-Kaplan Executive Function System battery (D-KEFS; Delis, Kaplan & Kramer, 2001) | Baseline, post-treatment (up to 20 weeks after baseline) and 12 months follow-up
  Measures executive function
Wisconsin Card Sorting Test: Computer Version 4 research edition (WCST-CV4; Heaton, PAR staff & Goldin 2003). | Baseline, post-treatment (up to 20 weeks after baseline) and 12 months follow-up
  Measures executive function
The California Verbal Learning Test (CVLT; Delis, Kramer & Kaplan, 1994). | Baseline, post-treatment (up to 20 weeks after baseline) and 12 months follow-up
  Measures memory
Wechsler Abbreviated Scale of Intelligence | Baseline
  Two subtests from Wechsler Abbreviated Scale of Intelligence (WASI; Wechsler, 1999) will be administered to assess IQ level.
Ambulatory Electrocardiogram (ECG) | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
  Measures heart rate variability (HRV)
Ekblom-Bak submaximal ergometer cycle test | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
  Test for prediction of VO2 max, which gives an indication of physical fitness
Strength test battery | Baseline, after pre-treatment (up to 8 weeks after baseline), post-treatment (up to 20 weeks after baseline), 6 months follow-up and 12 months follow-up
  Measures submaximal physical strength, which gives an indication of physical fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Hovland, PhD, Principal Investigator — Solli DPS, University of Bergen
Locations (1):
- Solli DPS, Bergen, Nesttun, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sirevag K, Stavestrand SH, Sjobo T, Endal TB, Nordahl HM, Andersson E, Nordhus IH, Rekdal A, Specht K, Hammar A, Halmoy A, Mohlman J, Hjelmervik H, Thayer JF, Hovland A. Physical exercise augmented cognitive behaviour therapy for older adults with generalised anxiety disorder (PEXACOG): a feasibility study for a randomized controlled trial. Biopsychosoc Med. 2023 Jul 19;17(1):25. doi: 10.1186/s13030-023-00280-7. PMID 37468978
- [Derived] Stavestrand SH, Sirevag K, Nordhus IH, Sjobo T, Endal TB, Nordahl HM, Specht K, Hammar A, Halmoy A, Martinsen EW, Andersson E, Hjelmervik H, Mohlman J, Thayer JF, Hovland A. Physical exercise augmented cognitive behaviour therapy for older adults with generalised anxiety disorder (PEXACOG): study protocol for a randomized controlled trial. Trials. 2019 Mar 18;20(1):174. doi: 10.1186/s13063-019-3268-9. PMID 30885256